CLINICAL TRIAL: NCT03272633
Title: Post-Transplant Use of Irradiated Haplo-Allogeneic Cells
Brief Title: Irradiated Donor Cells Following Stem Cell Transplant in Controlling Cancer in Patients With Hematologic Malignancies
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Roger Strair, MD, PhD, Professor of Medicine, RWJMS, Rutgers Cancer Institute of New Jersey
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 011702; NCI-2017-01537 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Pro20170000537; 011702 (Other: Rutgers Cancer Institute of New Jersey); P30CA072720 (NIH)
Record Dates: First submitted 2017-08-24; First posted 2017-09-05 (Actual); Results first posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia in Remission; Hematopoietic Cell Transplantation Recipient; JAK2 Gene Mutation; Loss of Chromosome 17p; Mantle Cell Lymphoma; Minimal Residual Disease; Myelodysplastic Syndrome; Non-Hodgkin Lymphoma; Plasma Cell Myeloma; RAS Family Gene Mutation; Recurrent Diffuse Large B-Cell Lymphoma; Recurrent Hematologic Malignancy; Recurrent Mature T- and NK-Cell Non-Hodgkin Lymphoma; Refractory Diffuse Large B-Cell Lymphoma; Refractory Mature T-Cell and NK-Cell Non-Hodgkin Lymphoma; Therapy-Related Acute Myeloid Leukemia; Therapy-Related Myelodysplastic Syndrome; TP53 Gene Mutation
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Chromosome 17 deletion; Lymphoma, Mantle-Cell; Neoplasm, Residual; Myelodysplastic Syndromes; Lymphoma, Non-Hodgkin; Multiple Myeloma; Lymphoma, Large B-Cell, Diffuse; Hematologic Neoplasms; Lymphoma, T-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort I (initial IHC within 42 days) (Experimental): Within 42 days after hematopoietic engraftment (both neutrophils and platelets) after autologous HSCT, patients receive initial treatment with IHC. Patients that do not have evidence of relapse or progressive disease may be treated every 8-12 weeks for up to 3 doses.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Biological: Irradiated Allogeneic Cells
- Cohort II (initial IHC within 70 days or after relapse) (Experimental): Patients with high-risk disease receive initial treatment with IHC within 70 days after hematopoietic engraftment (both neutrophils and platelets) after allogeneic HSCT. Patients being treated for relapsed disease may receive initial treatment with IHC any time after relapse is documented. Patients that do not have evidence of relapse or progressive disease may be treated every 8-12 weeks for up to 3 doses.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Biological: Irradiated Allogeneic Cells

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Receive IHC
  Other Names: Allogeneic Hematopoietic Cell Transplantation; allogeneic stem cell transplantation; HSC; HSCT
Biological: Irradiated Allogeneic Cells — Correlative studies

SUMMARY:
This pilot clinical trial studies the side effects of irradiated donor cells following stem cell transplant in controlling cancer in patients with hematologic malignancies. Transfusion of irradiated donor cells (immune cells) from relatives may cause the patient's cancer to decrease in size and may help control cancer in patients receiving a stem cell transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the toxicity associated with the administration of irradiated haploidentical cells (IHC) to patients with high-risk hematologic malignancies.

SECONDARY OBJECTIVES:

I. To determine if there is evidence of disease response associated with IHC.

TERTIARY OBJECTIVES:

I. To determine if treatment with the irradiated cells induces an immune response targeting tumor associated epitopes.

OUTLINE: Patients are assigned to 1 of 2 cohorts.

COHORT I: Within 42 days after hematopoietic engraftment (both neutrophils and platelets) after autologous hematopoietic stem cell transplantation (HSCT), patients receive initial treatment with IHC. Patients that do not have evidence of relapse or progressive disease may be treated every 8-12 weeks for up to 3 doses.

COHORT II: Patients with high-risk disease receive initial treatment with IHC within 70 days after hematopoietic engraftment (both neutrophils and platelets) after allogeneic HSCT. Patients being treated for relapsed disease may receive initial treatment with IHC any time after relapse is documented. Patients that do not have evidence of relapse or progressive disease may be treated every 8-12 weeks for up to 3 doses.

After completion of study treatment, patients will be followed up within 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patient with disease (stage) eligible per cohort
* COHORT 1: patients undergoing high dose chemotherapy with autologous stem cell rescue and ?high-risk? disease as defined below:

  * Diffuse large cell lymphoma or peripheral T cell lymphoma (including specified World Health Organization [WHO] subtypes) not in computed tomography (CT)-positron emission tomography (PET) complete remission at time of high dose therapy
  * Diffuse large cell lymphoma with ?double hit? or ?double expressor? features
  * Diffuse large cell lymphoma or peripheral T cell lymphoma (including WHO specified subtypes) refractory to standard induction therapy OR relapsing within 1 year of treatment OR in greater that second complete remission (CR)
  * Mantle cell lymphoma not in CR1
  * Multiple myeloma with ONE (or more) of the following high risk features:

    * Less than very good partial remission at time of high dose therapy
    * High Revised-International Staging System (R-ISS) (stage III ? 2 microglobulin >= 5.5 plus lactate dehydrogenase [LDH] > upper limit of normal [ULN] and/or del17p, t(4;14), t(14;16)) at time of diagnosis
    * Cytogenetics or fluorescent in situ hybridization (FISH) del17p
* COHORT 2: patients with high risk disease having undergone an allogeneic hematopoietic stem cell transplant from a 10/10 human leukocyte antigen (HLA) matched donor with one of the following disease subtypes:

  * Acute myeloid leukemia (AML) in CR1 with high risk features (European Leukemia Network [ELN]) at presentation

    * Diagnostic sample with either t(6;9), t(9;22), 11q23, inv 3, -5, -7, del17p, complex cytogenetics, NPMwt-flt3ITD+, OR p53 mutation (mut); patients whose samples have mutations in RUNX1 or ASXL1 are also eligible (unless the patient has favorable cytogenetics)
  * AML in CR1 with measurable minimal residual disease (MRD) by molecular (e.g., myeloid mutation profile, polymerase chain reaction [PCR] for NPM1, core-binding factor [CBF], mixed lineage leukemia [MLL]) or flow cytometry
  * AML not in CR1 (including patients with morphologic CR but with incomplete recovery, CRi)
  * Myelodysplastic syndrome (MDS) with complex cytogenetics, 17p deletion or p53 mutation, or JAK2 or RAS mutation
  * Treatment-related MDS or AML
  * Acute lymphoblastic leukemia (ALL) not in CR1
  * ALL with MRD
  * Any hematologic malignancy relapsed or with persistent disease after allogeneic hematopoietic stem cell transplant
  * Multiple myeloma
  * Non-Hodgkin lymphoma (NHL) with chemoresistant disease at time of transplant
  * Any patient undergoing allogeneic hematopoietic stem cell transplant and an anticipated rate of relapse > 80% based upon published data and for which there is consensus amongst the Hematologic Malignancies Tumor Study Group that enrollment is appropriate
* Availability of a genetic child, genetic parent or sibling as a potential HLA haploidentical donor
* Meets standard eligibility requirements for high dose chemotherapy with autologous stem cell rescue (COHORT 1) or allogeneic hematopoietic stem cell transplant (COHORT 2) and has signed consent for those procedures
* DONOR: Donor must be related to patient and be partially (>= 3/6 antigen) HLA-matched
* DONOR: Donor must meet all Robert Wood Johnson (RWJ) Blood Services requirements for hematopoietic stem cell donation including:

  * Age >= 18 years old;
  * Normal hemogram (white blood cells [WBC] 4.0-10.0 x 10^3/mm^3; platelet count 150,000 to 440,000/mm^3 ; hemoglobin/hematocrit; 12.5-18 g/dl, 38 to 54%
  * Not pregnant or lactating;
  * Not human immunodeficiency virus (HIV)-1, HIV-2, hepatitis C virus (HCV), hepatitis B core or human T-cell lymphotropic virus (HTLV)-I/II seropositive; hepatitis B surface antigen (HB S ag) (-); meet other infectious disease screening criteria utilized by RWJ Blood Services;
  * No uncontrolled infections, other medical or psychological/social conditions, or medications that might increase the likelihood of patient or donor adverse effects or poor outcomes;
  * Meet other blood bank criteria for blood product donation (as determined by RWJ Blood Center screening history and laboratory studies)

Exclusion Criteria:

* Non-English speaking person
* Patients undergoing haploidentical allogeneic hematopoietic stem cell transplants are not eligible; patients undergoing < 10/10 HLA allele matched allogeneic transplant are not eligible
* Pregnant women
* DONOR: Non-English speaking person
* DONOR: Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Strair, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort I (Initial IHC Within 42 Days) | Cohort II (Initial IHC Within 70 Days or After Relapse)
Started | 0 | 2
Completed | 0 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants qualified for cohort I
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort I (Initial IHC Within 42 Days) | Cohort II (Initial IHC Within 70 Days or After Relapse) | Total
Number analyzed (Participants) | 0 | 2 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 2 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Received Irradiated Haploidentical Cells (IHC) With Disease Response
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Up to 8 weeks after last protocol treatment
Population: no data was collected. Refers to the Cohort 1 Arm
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort I (Initial IHC Within 42 Days) | Cohort II (Initial IHC Within 70 Days or After Relapse)
Number analyzed (Participants) | 0 | 2
Participants |  | 2

2. Primary Outcome: the Number of Participants With Toxicities Associated With Administration of Irradiated Haploidentical Cells (IHC) Evaluated According to Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
Description: The anticipated/projected IHC-associated toxicities of greatest concern include: short-term toxicities- constitutional/systemic adverse events including fevers, hypotension, pulmonary infiltrates; long-term toxicities: autoimmune effects, graft-versus-host disease (GVHD), graft rejection. Toxicity will be measured by occurrence of any experimental treatment-related adverse events (AE) up to 12 weeks of completion of therapy. The CTCAE version 4.0 will be utilized for the description and grading of the AE. All symptoms, signs, or diseases assessed as experimental treatment-related will be captu
Time Frame: Up to 12 weeks of completion of therapy
Population: no data was collected. Refers to the Cohort 1 Arm
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort I (Initial IHC Within 42 Days) | Cohort II (Initial IHC Within 70 Days or After Relapse)
Number analyzed (Participants) | 0 | 2
Participants |  | 2

3. Secondary Outcome: Induction of Host T Cells Reactive With Tumor Associated Epitopes
Description: It will be determined if treatment with the irradiated cells induces an immune response targeting tumor associated epitopes.
Time Frame: Up to 8 weeks after last protocol treatment
Population: no data was collected
Arm/Group | Cohort I (Initial IHC Within 42 Days) | Cohort II (Initial IHC Within 70 Days or After Relapse)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 8 weeks after last protocol treatment
Description: no data was collected. Adverse Events Description text only refers to the Cohort II No participants were enrolled in Cohort I, so no adverse events were monitored/assessed for Cohort I
Arm/Group | Cohort I (Initial IHC Within 42 Days) | Cohort II (Initial IHC Within 70 Days or After Relapse)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/2
Other Adverse Events (participants affected / at risk) | 0/0 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort I (Initial IHC Within 42 Days) (N=0) | Cohort II (Initial IHC Within 70 Days or After Relapse) (N=2)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort I (Initial IHC Within 42 Days) (N=0) | Cohort II (Initial IHC Within 70 Days or After Relapse) (N=2)
General disorders and administration site conditions (General disorders) | 0 (0) | 2
Investigations (Investigations) | 0 (0) | 2 (5)
Eye disorders (Eye disorders) | 0 (0) | 1 (1)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Nervous system disorders (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-23): https://cdn.clinicaltrials.gov/large-docs/33/NCT03272633/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-23): https://cdn.clinicaltrials.gov/large-docs/33/NCT03272633/ICF_001.pdf